CLINICAL TRIAL: NCT01823809
Title: Assessment of Coronary Artery Disease With Multi-Slice Computed Tomography Combined With Stress Cardiac Magnetic Resonance Imaging Compared to Coronary Angiography Combined With Fractional Flow Reserve Trial
Brief Title: Non-invasive and Invasive Assessment of Coronary Artery Disease
Acronym: COMFORT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Problems with inclusion, >80% of patients included
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Gabija Pundziute, Principal Investigator, University Medical Center Groningen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: METc2011.084
Record Dates: First submitted 2013-03-04; First posted 2013-04-04 (Estimated); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease; Computed Tomography; Cardiac Magnetic Resonance; Fractional Flow Reserve
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Imaging arm (Other): There is one study arm only. The imaging modalities will be performed in all patients.
  Interventions: Device: adenosine stress Cardiac Magnetic Resonance Imaging

INTERVENTIONS:
Device: adenosine stress Cardiac Magnetic Resonance Imaging

SUMMARY:
The purpose of the study is to assess the diagnostic accuracy of a combined use of non-invasive coronary angiography with multi-slice computed tomography (MSCT) and stress cardiac magnetic resonance (CMR) imaging in patients with obstructive lesions on MSCT and with low to intermediate pre-test likelihood of coronary artery disease (CAD) as compared to invasive coronary angiography (CAG) and Fractional Flow Reserve (FFR) measurements.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with stable angina pectoris with low to intermediate pre-test likelihood of CAD;
2. no previous history of CAD;
3. obstructive stenosis (≥50% luminal narrowing) on MSCT coronary angiography; 4.informed consent.

Exclusion Criteria:

1. patients with a previous history of CAD;
2. patients with contraindications for MSCT: a.cardiac rhythms other than sinus rhythm, b.pregnancy, c.allergy for contrast medium, d.renal failure (estimated glomerular filtration rate (eGFR) < 50ml/min), e.resting heart rate >75 bpm plus contra-indications for beta-blockade, f. weight >100 kilograms;
3. contraindications for cardiac magnetic resonance (CMR) imaging: a.MR-incompatible implants, b. Claustrophobia, c. contraindications for adenosine: i. known or suspected hypersensitivity to adenosine, ii. known or suspected bronchoconstrictive or bronchospastic disease, iii. 2nd or 3rd degree atrioventricular (AV) block, iv. Sinus bradycardia (heart rate < 45 bpm), v. Systemic arterial hypotension (<90 mmHg). d. contraindications for gadolinium: i. renal failure (estimated eGFR <30 ml/min);
4. no informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2011-11 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy to detect ischemia with stress CMR compared to FFR | one month
  The diagnostic accuracy of MSCT coronary angiography in combination with stress CMR imaging as compared to invasive CAG and FFR measurement, as a standard of reference to detect obstructive and hemodynamically significant stenoses in patients with low to intermediate pre-test likelihood of CAD.

SECONDARY OUTCOMES:
Predictive value for treatment strategy of a non-invasive strategy with MSCT and stress CMR compared to an invasive strategy | one month
  to evaluate whether MSCT coronary angiography in combination with stress CMR imaging may accurately predict treatment strategy (medical therapy versus revascularization therapy) as compared to CAG and FFR in patients with low to intermediate pre-test likelihood of CAD.

CONTACTS AND LOCATIONS:
Overall Officials: Gabija Pundziute, MD, PhD, Principal Investigator — University Medical Center Groningen, Department of Cardiology
Locations (2):
- University Medical Center Groningen, Departments of Cardiology and Radiology, Groningen, Netherlands
- University Hospital Linköping, Departments of Clinical Physiology, Cardiology and Center for Medial Imaging Visualization, Linköping, Sweden